CLINICAL TRIAL: NCT04475315
Title: Left Ventricular Papillary Muscle Sling for Heart Failure With Reduced Ejection Fraction (Papillary Muscle Sling)
Brief Title: Ventricular Sling for Heart Failure With Reduced Ejection Fraction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Lamelas, Chief and Program Director of Cardiothoracic Surgery, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200679
Record Dates: First submitted 2020-07-10; First posted 2020-07-17 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure; Cardiomyopathy, Dilated
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Papillary Muscle Sling Group (Experimental): Participants in the papillary muscle sling group will receive the sling technique performed in conjunction with their standard of care (SOC) Coronary Artery Bypass Grafting (CABG) surgery.
  Interventions: Device: Papillary Muscle Sling; Procedure: CABG surgery
- Controls Group (Active Comparator): Participants in the control group will receive their SOC CABG surgery only, without any additional intervention.
  Interventions: Procedure: CABG surgery

INTERVENTIONS:
Device: Papillary Muscle Sling — The sling is made of a Gore-Tex sheet or by using a 4 mm Gore-Tex vascular graft implanted around the base of the papillary muscles and tightened.
  Arms: Papillary Muscle Sling Group
Procedure: CABG surgery — Standard of care Coronary Artery Bypass Grafting (CABG) surgery will be performed to improve blood flow to the heart by bypassing the narrowed segment of a severely diseased coronary artery

SUMMARY:
The purpose of this research is to investigate the effect of using this surgical technique in conjunction with bypass surgery to improve heart function and size, as well as decrease the possibility of future mitral valve surgery.

DETAILED DESCRIPTION:
The Sling is used to draw together the ventricular walls at the base of the papillary muscles. This technique has previously been used in conjunction with mitral valve surgery, and has shown significant benefits for the patients.

The reduction in the lateral inter-papillary muscle separation and in the left ventricular volume provided by this technique is expected to improve ventricular function, limit progression of ventricular dilation, and avoid progression of MR when performed without mitral valve surgery in patients with symptomatic ventricular dilation.

ELIGIBILITY:
Inclusion Criteria:

Patients with symptomatic heart failure with reduced ejection fraction and either ischemic or non-ischemic cardiomyopathies, referred for CABG surgery. Suitability for the ventricular sling procedure is determined by the surgeon and or cardiologist, using some or all the criteria described below:

* Left ventricular end diastolic diameter is greater than or equal to 55mm.
* Ejection fraction ≥20% and ≤40%
* FMR grade ≤ 2+ (≤ mild FMR) as defined by the guidelines of the American society of echocardiography at the time of the study approval (via a transthoracic or transesophageal echo).
* End-systolic Interpapillary muscle distance ≥ 20mm
* Cardiomyopathy of ischemic or non-ischemic origins.
* Able to sign informed consent and release of medical information forms, or able to assign a legal representative who can sign on the patient's behalf.

Exclusion Criteria:

* Any evidence of structural (chordal or leaflet) mitral lesions.
* Planned concomitant intra-operative procedures (except for closure of patent foramen ovale or atrial septal defect or coronary revascularization)
* Planned concomitant intra-operative Maze procedure for symptomatic paroxysmal atrial fibrillation.
* Persistent atrial fibrillation
* Prior mitral valve repair
* Contraindication for cardiopulmonary bypass
* Clinical signs of cardiogenic shock
* ST segment elevation myocardial infarction within 14 days prior to inclusion in this study.
* Congenital heart disease (except PFO or ASD)
* Chronic renal insufficiency defined by Creatinine ≥ 3.0 or chronic renal replacement therapy, who are contraindicated for cardiac surgery
* Recent history of psychiatric disease that is likely to impair compliance with the study protocol, in the judgement of the investigator
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular function as assessed by LVEF | Baseline, up to 5 years
  Change in Left Ventricular Ejection Fraction (LVEF) will be reported as a change in percent ejection fraction assessed via echocardiogram
Change in left ventricular volume | Baseline, up to 5 years
  End systolic and end diastolic left ventricular volumes will both be evaluated in mL using echocardiogram.

SECONDARY OUTCOMES:
Mortality Rate | 5 years
  Rate of reported mortality rate will be evaluated.
Number of Major Adverse Cardiac Events (MACE) | 5 years
  MACE is defined as a composite of clinical events comprised of death, stroke, worsening heart failure defined as +1 New York Heart Association (NYHA) class, Congestive Heart Failure (CHF) hospitalization and mitral valve intervention as evaluated by treating physician
Percentage of participants at each FMR severity grade | Baseline, up to 5 years
  Functional Mitral Regurgitation (FMR) severity is graded on a scale of 1 to 4 with 1 = none, 2 =mild, 3 = moderate and 4 =severe. This outcome will report the percentage of participants with reported none, mild, moderate or severe mitral regurgitation as assessed via echocardiogram by treating physician.
Change in MLHF Questionnaire Score | Baseline, up to 5 years
  Minnesota Living with Heart Failure (MLHF) is a 21-item questionnaire with a total score ranging from 0 (indicating heart failure has no affect to life) to 105 (indicating the greatest affect to life).
Change in Functional Status as assessed by 6MWT | Baseline, up to 5 years
  Functional status will be assessed as the distance reached in meters via the 6-minute Walk Test (6MWT).
All Cause Readmission Rate | 5 years
  All cause readmission rate will be calculated for any case throughout the duration of study participation.
Heart Failure Readmission Rate | 5 years
  Heart failure readmission rate will be calculated for heart failure throughout the duration of study participation.
Incidence of Mitral Leaflet Tenting | 5 years
  Mitral Leaflet tenting will be evaluated using echocardiographic imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Lamelas, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamelas J, Mihos C, Santana O. Surgical technique: papillary muscle sling for functional mitral regurgitation during minimally invasive valve surgery. Heart Surg Forum. 2013 Oct;16(5):E295-7. doi: 10.1532/hsf98.2013209. PMID 24364086
- [Background] Santana O, Solenkova NV, Pineda AM, Mihos CG, Lamelas J. Minimally invasive papillary muscle sling placement during mitral valve repair in patients with functional mitral regurgitation. J Thorac Cardiovasc Surg. 2014 Jan;147(1):496-9. doi: 10.1016/j.jtcvs.2013.03.006. Epub 2013 Mar 29. PMID 23545430